CLINICAL TRIAL: NCT06940843
Title: Enhancing Social Connection, Health, and Aging in Older Persons: A Pilot Randomized Trial of the Hopeful and Healthy Living (HHL) Program
Brief Title: A Pilot Randomized Controlled Trial of the Hopeful and Healthy Living Program
Acronym: (HHL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Bay Cove Human Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7458B; 90RTHF0007 (Other Grant/Funding Number: Nat. Ins. on Disability, Indepen. Living and Rehab Research)
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Serious Mental Illness; Older Adults
Keywords: psychosocial interventions; cognitive interventions; social skills interventions; healthy lifestyle interventions; older adults with SMI

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HHL group participants (Experimental): Participants will complete the 16-week manualized HHL intervention. This group intervention will occur weekly for 90 minutes. These participants will also continue with treatment as usual.
  Interventions: Behavioral: Hopeful and Healthy Living (HHL)
- Treatment as usual (No Intervention): Participants assigned to this arm will continue with treatment as usual.

INTERVENTIONS:
Behavioral: Hopeful and Healthy Living (HHL) — The HHL intervention is a 16-week long, manualized group intervention. Classes will be held weekly for 90 minutes. The class covers 15 topics centered on building social connections, developing healthy lifestyle routines around eating, exercise, and sleep. Each class will target one social skill (i.e. starting conversations) and one cognitive self-management strategy (i.e. memory tips), which will be taught and practiced in class. Each class also includes a facilitated exercise component and individually tailored take home application activity.
  Arms: HHL group participants

SUMMARY:
The goal of this clinical trial is to learn if a novel psychosocial intervention is effective in helping adults over 50 with serious mental illness (SMI) increase their social connections and participate in more healthy lifestyle activities. The Hopeful and Healthy Living (HHL) intervention combines social skills training and training in cognitive self-management strategies in order to help older adults build healthy lifestyle and social routines. We predict that:

* Individuals who participate in the HHL intervention will improve more in perceived social support (i.e., what people get from relationships such as reliance, reassurance of worth, attachment) and loneliness at the 4-, 8-, and 12-month follow-up assessments than those who receive treatment as usual (TAU).
* Individuals who participate in the HHL intervention will improve more in overall psychosocial functioning at the 4-, 8-, and 12-month follow-up assessments than those who receive TAU.
* Individuals who participate in the HHL intervention will improve more in cognitive functioning at the 4-, 8-, and 12-month follow-up assessments than those who receive TAU.
* Individuals who participate in the HHL intervention will improve more in healthy behaviors (sleep, activity, diet) at the 4-, 8-, and 12-month follow-up assessments than those who receive TAU.

In this trial, participants will be either receive the HHL intervention or participate in their regular treatment activities (treatment as usual). HHL vs. TAU will be compared to see if there are any differences in social support, cognition, loneliness, psychosocial functioning, or healthy lifestyle activities including physical activity, sleep, and diet.

Participants will be asked to complete an interview-based assessment at baseline, 4-months, 8-months, and 12-months. After completing the baseline assessment, those who are in the experimental group will participate in the 16-week long HHL group intervention.

ELIGIBILITY:
Inclusion Criteria:

50 years or older, diagnosis of a serious mental illness, and a member of Center Club or Transitions of Boston

Exclusion Criteria:

Diagnosis of dementia or other progressive neurological disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | Baseline, 4-, 8-, 12- month followup
  Standardized screening tool used for assessing cognition.
The Cognitive Self-Efficacy Scale | Baseline, 4-, 8-, 12- month followup
  10-item measure that assesses confidence in everyday cognitive tasks.
The DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure | Baseline, 4-, 8-, 12- month followup
  Adult will be used to assess and statistically control for mental health symptom severity.
The UCLA Loneliness Scale-3-item instrument | Baseline, 4-, 8-, 12- month followup
  3-item screening tool for loneliness.
The Social Provisions Scale | Baseline, 4-, 8-, 12- month followup
  24-item instrument that will be used to measure various types of social supports.
The Physical Activity Scale for the Elderly (PASE) | Baseline, 4-, 8-, 12- month followup
  Standardized measurement of physical activity related to exercise, work, recreation, and daily living activities.
Starting the Conversation | Baseline, 4-, 8-, 12- month followup
  A brief standardized survey for assessing daily eating habits.
Pittsburg Sleep Quality Index (PSQI) | Baseline, 4-, 8-, 12- month followup
  An 11-item tool that is used to assess sleep quality and routines.

SECONDARY OUTCOMES:
HHL Group Satisfaction and Feedback Survey | 4-month assessment only
  For experimental group participants only.

CONTACTS AND LOCATIONS:
Overall Officials: Susan McGurk, PhD, Principal Investigator — Boston University; Kim Mueser, PhD, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Bay Cove Center Club, Boston, Massachusetts
  - Bay Cove Transitions of Boston, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No